CLINICAL TRIAL: NCT04163003
Title: Targeted Intervention for Insufficient Sleep Among Typically-Developing Adolescents
Acronym: TAPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jessica Levenson, Assistant Professor of Psychiatry and Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19080033; K23HD087433 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-11-14 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: Among those with insufficient sleep, after participants are screened and receive universal education about sleep, those with insufficient sleep will be offered to participate in the randomized pilot trial. There are two arms in the randomized trial: TAPAS intervention, and wait-list control (monitoring only). The study will enroll n=50 participants in the Randomized Control Trial (RCT) to obtain full data on n=40 participants after attrition.
  Participants who obtain sufficient sleep will not be randomized, but will obtain the universal education only. Investigators anticipate enrolling n=35 adolescents with sufficient sleep.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAPAS (Experimental): Participants will participate in the TAPAS intervention, which will consist of one in-person engagement session with a therapist and 8 weeks of web-based automated intervention prompts. The program will utilize empirically supported approaches for promoting sleep health, delivered in-person and via text-message, focusing on: tailored psychoeducation, motivation and efficacy to change sleep, extending sleep duration, and regularizing sleep timing across the week.
  Interventions: Behavioral: Targeted Approaches for Promoting Adolescent Sleep (TAPAS)
- Sleep monitoring only, then TAPAS (Experimental): Participants will participate in sleep monitoring only first, then participate in the TAPAS intervention. First, participants will monitor sleep with sleep diary, but they will not receive feedback or any other information on to sleep.TAPAS will consist of one engagement session with a therapist and 4 weeks of web-based automated intervention prompts. The program will utilize empirically supported approaches for promoting sleep health, delivered in-person and via text-message, focusing on: tailored psychoeducation, motivation and efficacy to change sleep, extending sleep duration, and regularizing sleep timing across the week. Sleep monitoring is proposed to last the same duration as the targeted intervention in this arm.
  Interventions: Behavioral: Targeted Approaches for Promoting Adolescent Sleep (TAPAS); Behavioral: Sleep Monitoring Only

INTERVENTIONS:
Behavioral: Targeted Approaches for Promoting Adolescent Sleep (TAPAS) — The targeted intervention is a three part sleep program, involving a 2- minute psychoeducation video, an in-person session with a clinician focusing on sleep, and web-based goal setting related to sleep behaviors. Intervention approaches to promoting adolescent sleep and reducing insufficient sleep use a motivational interviewing style, rooted in cognitive-behavioral strategies for improving sleep.
  Other Names: TAPAS
Behavioral: Sleep Monitoring Only — Participants will monitor sleep with sleep diary, but they will not receive feedback or any other information on to sleep.
  Arms: Sleep monitoring only, then TAPAS

SUMMARY:
The overall aim of Dr. Levenson's research proposal is to test the acceptability, feasibility, and preliminary outcomes of a sleep promotion program delivered to 13-15 year olds who report insufficient sleep. Dr. Levenson will examine the feasibility and acceptability of the program through a randomized pilot trial (n=40) that uses a two-period, wait-list control design. Then, Dr. Levenson will test whether the program is associated with changes in sleep, motivation, and four outcome domains: academic functioning, attention, risk behavior, and affect. Such a broadly relevant program has the potential for enormous public health impact by improving sleep and facilitating healthy development across a range of domains among typically-developing adolescents who are highly vulnerable to adverse consequences.

DETAILED DESCRIPTION:
General Description:

This study has two sub-studies: one for youth who experience behaviorally insufficient sleep syndrome (BISS) and one for youth who obtain sufficient sleep. This includes a randomized controlled trial for youth who obtain insufficient sleep (BISS), and a universal education (UE) only intervention for youth who obtain sufficient sleep.

All participants will complete a pre-consent screen. Those with sufficient sleep will complete consent/assent and a full screening assessment, and they will watch a sleep education video (UE). If eligible for the sufficient sleeper study, the full screening assessment will serve as a baseline assessment as well. Participants will complete a follow-up assessment about one month later.

Those who pre-screen as insufficient sleepers will complete consent/assent, complete a full screening process, and watch a sleep education video (UE). Those who remain eligible after the full screening process will complete a baseline assessment. Then, youth will be randomized to the TAPAS intervention or to a wait-list control (monitoring only). After completing the post-period 1 follow-up assessment, those in the wait-list control group will switch to the other arm, via a cross-over design. Participants in the intervention-first group will continue to receive the intervention iin Period 2 after post-period 1. After this period, participants will complete the post-period 2 follow-up assessment.

Detailed Description:

Participants. Youth ages 13-15 will be recruited through various methods (e.g., social media advertising, University research registry, flyers, email listservs and online magazines, and from the waiting room of the Children's Hospital of Pittsburgh Center for Adolescent and Young Adult Health (CAYAH)). Among those screened, the investigators will deliver universal education about sleep and conduct baseline and follow-up assessments among n=35 sufficient sleepers. Investigators will randomize n=50 with insufficient sleep to the TAPAS intervention or wait-list control (monitoring only). Overall, investigators plan to collect complete data on n=40 participants, after attrition.

Baseline assessments will include: measures of sleep (sleep diary and actigraphy), academic functioning, attention, affect, motivation, and risk behavior.

TAPAS Intervention. Program goals are to increase knowledge about healthy sleep practices, to increase sleep duration by going to bed earlier (sleep extension), and to increase regularity in sleep timing over the week by limiting oversleeping on the weekends. During the 45-60 minute intervention session, the youth and clinician will discuss the youth's sleep timing and quality and explore the youth's attitudes and social influences on sleep. The clinician will develop discrepancies between current sleep behavior and the youth's values and goals.

It is proposed that the 4-8-week text messaging/web-based portion of the intervention will begin immediately after the clinician session. Participants will receive twice-weekly summaries of their sleep based on diary entries. Participants will then be asked via the web if they'd like to modify their sleep, providing them with autonomy in their answer. Investigators will rely on strategies for extending and regularizing sleep.

Wait-List Control (monitoring only) Condition. The wait-list is proposed to last half the duration as the targeted intervention (4 vs 8 weeks). Participants will monitor sleep with the sleep diary, but they will not receive feedback or any other information on their sleep.

Participants will repeat the baseline assessments and 7 days of actigraphy at the end of Period 1 and at the end of Period 2 (only those randomized to Wait-List Control will cross-over to TAPAS intervention for Period 2).

Follow-up assessments will include: measures of sleep (sleep diary and actigraphy), academic functioning, attention, affect, motivation, and risk behavior.

ELIGIBILITY:
All participants will be excluded if they live more than roughly an hour's drive from Pittsburgh, Pennsylvania (PA).

Insufficient Sleepers:

Investigators will screen, deliver universal education (UE), and offer participation to all participants:

1. ages 13 years, 0 months to 15 years, 11 months;
2. able and willing to give informed assent to participate (with informed consent from parent);
3. insufficient sleep (≤7.5 hours sleep on average weeknights); and
4. weekend-weekday sleep timing shift >=1.5 hours.

Inclusion criteria are not applicable for parents.

Exclusion Criteria:

1. Evidence of mental retardation, pervasive developmental disorder, or organic central nervous system disorder will exclude potential participants;
2. unstable medical conditions;
3. use of psychotropic medications or medications known to impact sleep;
4. adolescent pregnancy;
5. clinical levels of psychopathology, except for youth with a sole diagnosis of gender dysphoria;
6. current sleep disorders except for sleep-onset insomnia;
7. extreme evening preference; and
8. Currently living >1 hour outside of the greater Pittsburgh region.

Sufficient Sleepers:

Inclusion Criteria:

1. ages 13-15;
2. sufficient sleep (>7.5 hours of sleep);
3. willing/able to provide informed assent/consent.

Exclusion Criteria:

1. Evidence of mental retardation, pervasive developmental disorder, or organic central nervous system disorder;
2. unstable medical conditions;
3. use of psychotropic medications or medications known to impact sleep;
4. adolescent pregnancy;
5. clinical levels of psychopathology, except for youth with a sole diagnosis of gender dysphoria;
6. current sleep disorders except for sleep-onset insomnia;
7. extreme evening preference; and
8. Currently living >1 hour outside of the greater Pittsburgh region.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Attrition | 4 weeks
  Participant attrition rate
Response Rate | 4 weeks
  Participant response rate to electronic intervention prompts
Adherence | 1 session
  A locally-developed Sleep Promotion Program Rating form indicates which program components covered in each clinician session. The measure is a checklist that indicates the presence or absence of each component covered in the session.
Participant Satisfaction | 4 weeks
  A locally-developed Treatment Satisfaction Questionnaire measures program satisfaction. Scores range from 18 to 75, with higher scores indicating greater satisfaction.
Sleep Diary Sleep Duration | 4 weeks
  Average sleep duration (in hours and minutes) as measured by sleep diary
Sleep Diary Sleep Timing | 4 weeks
  Average sleep timing as measured by sleep diary
Sleep Diary Weekend-Weekday Sleep Timing Differences | 4 weeks
  Difference in average weekend and weekday sleep timing as measured by sleep diary

SECONDARY OUTCOMES:
Actigraphy Sleep Duration | 4 weeks
  Average sleep duration (in hours and minutes) as measured by actigraphy
Actigraphy Sleep Timing | 4 weeks
  Average sleep timing as measured by actigraphy
Actigraphy Weekend-Weekday Sleep Timing Differences | 4 weeks
  Differences in average weekend and weekday sleep timing as measured by actigraphy

OTHER OUTCOMES:
Academic Functioning | 4 weeks
  Grades in School
Attention | 4 weeks
  The Psychomotor Vigilance Test (PVT) is a computer-based test of vigilant attention, which is measured by reaction time in milliseconds.
Affect | 4 weeks
  The Mood and Feelings Questionnaire (MFQ) is a measure or depressive symptoms. Scores range from 0 to 66, with higher scores indicating greater depressive symptoms.
Risk Behavior | 4 weeks
  The Balloon Analogue Risk Task (BART) is a computerized measure of risk-taking behavior. In the task, the participant can earn money by pumping up balloons. Each pump incrementally results in a larger balloon and an associated increase in earn money. However, popping a balloon results in loss of money. Each balloon pops at a different point. The primary outcome is average number of pumps on unexploded balloons, with higher scores indicative of greater risk-taking propensity

CONTACTS AND LOCATIONS:
Overall Officials: Jessica C Levenson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wescott DL, Goldstein TR, Wallace ML, Miller E, Buysse DJ, Harvey A, Suffoletto B, Rofey DL, Levenson JC. Effects of a single session intervention on actigraphy-measured sleep for adolescents with insufficient and irregular sleep: A randomized controlled trial. Sleep Health. 2026 Jan 19:S2352-7218(25)00280-3. doi: 10.1016/j.sleh.2025.12.008. Online ahead of print. PMID 41558877
- [Derived] Levenson JC, Goldstein TR, Wallace ML, Witt R, Harvey AG, Buysse D, Rofey DL, Suffoletto B, Miller E. A sleep promotion program for insufficient sleep among adolescents: a pilot feasibility randomized controlled trial. J Clin Sleep Med. 2025 Mar 1;21(3):529-541. doi: 10.5664/jcsm.11456. PMID 39506293